CLINICAL TRIAL: NCT06660173
Title: A Study to Evaluate the Efficacy, Safety & Tolerability of Maridebart Cafraglutide in Adults With T2DM
Brief Title: A Study of Maridebart Cafraglutide in Adult Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230143; 2024-513539-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Obesity; AMG 133; T2DM; Hemoglobin A1C (HbA1c)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide (Experimental): Participants will be randomized to receive maridebart cafraglutide at varying dose levels, or placebo, for up to 24 weeks. Participants who complete the 24-week Part 1 treatment period and meet specific criteria will have the option to begin an exploratory part 2 where they will be re-randomized to receive maridebart cafraglutide for an additional 24 weeks. Participants who complete the 24-week Part 2 treatment period and meet specific criteria will have the option to begin an exploratory part 3 where they will be re-randomized to receive maridebart cafraglutide for an additional 24 weeks.
  Interventions: Drug: Maridebart Cafraglutide
- Placebo (Placebo Comparator): Participants will be randomized to receive maridebart cafraglutide at varying dose levels, or placebo, for up to 24 weeks. Participants who complete the 24-week Part 1 treatment period and meet specific criteria will have the option to begin an exploratory part 2 where they will be re-randomized to receive maridebart cafraglutide for an additional 24 weeks. Participants who complete the 24-week Part 2 treatment period and meet specific criteria will have the option to begin an exploratory part 3 where they will be re-randomized to receive maridebart cafraglutide for an additional 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Solution for subcutaneous injection.
  Other Names: AMG 133
  Arms: Maridebart Cafraglutide
Drug: Placebo — Solution for subcutaneous injection.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the dose-response relationship of maridebart cafraglutide on glucose control compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening (or ≥ legal age within the country if it is older than 18 years)
* Type 2 diabetes for ≥6 months according to the World Health Organization classification
* HbA1c of 7.0% to 10.5%, inclusive, as assessed by the central laboratory
* Treatment of diabetes with diet and exercise alone, or with a stable dose of metformin, with or without a sodium-glucose cotransporter-2 inhibitor, for at least 3 months prior to screening
* Body mass index of 23 to 50 kilograms per square meter

Exclusion Criteria:

* Type 1 diabetes
* Use of any glucose-lowering medication, other than metformin with or without a sodium-glucose cotransporter-2 inhibitor, within 3 months prior to screening
* Estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 square meter, calculated by the Chronic Kidney Disease-Epidemiology equation.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy
* History of acute or chronic pancreatitis
* Malignancy within 5 years before screening, except for nonmelanoma skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer
* Myocardial infarction, unstable angina, coronary artery bypass graft surgery or other major cardiovascular surgery, percutaneous coronary intervention, transient ischemic attack, cerebrovascular accident, or decompensated congestive heart failure within 90 days prior to screening, or currently have New York Heart Association Class III or IV heart failure.
* Use of medications that affect glucose control or body weight or history of bariatric surgery or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 24 in Hemoglobin A1c (HbA1c) | Baseline to Week 24

SECONDARY OUTCOMES:
Percent Change From Baseline to Week 24 in Body Weight | Baseline to Week 24
Number of Participants Achieving HbA1c < 7.0% at Week 24 | Week 24
Number of Participants Achieving HbA1c ≤ 6.5% at Week 24 | Week 24
Number of Participants Achieving ≥ 5% Reduction in Body Weight From Baseline at Week 24 | Week 24
Number of Participants Achieving ≥ 10% Reduction in Body Weight From Baseline at Week 24 | Week 24
Change From Baseline to Week 24 in Fasting Glucose | Baseline to Week 24
Percent Change From Baseline to Week 24 in Total Cholesterol | Baseline to Week 24
Percent Change From Baseline to Week 24 in Low-density Lipoprotein Cholesterol (LDL-C) | Baseline to Week 24
Percent Change From Baseline to Week 24 in High-density Lipoprotein Cholesterol (HDL-C) | Baseline to Week 24
Percent Change From Baseline to Week 24 in Non-high Density Lipoprotein Cholesterol (non-HDL-C) | Baseline to Week 24
Percent Change From Baseline to Week 24 in Very-low-density Lipoprotein Cholesterol (VLDL-C) | Baseline to Week 24
Percent Change From Baseline to Week 24 in Triglycerides | Baseline to Week 24
Percent Change From Baseline to Week 24 in Free Fatty Acids (FFA) | Baseline and Week 24
Change From Baseline to Week 24 in Systolic Blood Pressure | Baseline and Week 24
Change From Baseline to Week 24 in Diastolic Blood Pressure | Baseline and Week 24
Change from Baseline to Week 24 in High-sensitivity C-reactive Protein | Baseline and Week 24
Pre-dose Plasma Concentration of Maridebart Cafraglutide at Week 20 | Week 20
Maximum Observed Plasma Concentration of Maridebart Cafraglutide at Week 20 | Week 20
Number of Participants with Treatment Emergent Adverse Events | Up to 24 Weeks
Number of Participants with Serious Adverse Events | Up to 24 Weeks
Number of Participants with Anti-maridebart Cafraglutide Antibody Formation | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (96):
- United States (28):
  - Accel Research Site - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - Hope Clinical Research LLC, Canoga Park, California
  - Orange County Research Center, Lake Forest, California
  - San Jose Clinical Trials, San Jose, California
  - Northeast Research Institute - Neri, Fleming Island, Florida
  - New Horizon Research Center, Miami, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Conquest Research - Winter Park, Winter Park, Florida
  - Accel Research Site - Neurostudies, Decatur, Georgia
  - Cedar Crosse Research and Health Care, Chicago, Illinois
  - Tandem Clinical Research - Marrero, Marrero, Louisiana
  - DM Clinical - Detroit, Southfield, Michigan
  - Montana Medical Research, Missoula, Montana
  - Physicians East, Greenville, North Carolina
  - Diabetes and Endocrinology Associates of Stark County Inc, Canton, Ohio
  - Alliance for Multispecialty Research, Norman, Oklahoma
  - Trial Management Associates - Myrtle Beach, Myrtle Beach, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - DM Clinical Research - Cyfair Clinical Research Center, Houston, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - DM Clinical Research - Martin Diagnostic Clinic, Tomball, Texas
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Manassas Clinical Research Center Inc, Manassas, Virginia
  - Eastside Research Associates Health Research, Redmond, Washington
- Austria (4):
  - Medizinische Universitaet Graz, Graz
  - Krankenhaus der Barmherzigen Brueder Linz, Linz
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Greece (6):
  - Laiko General Hospital of Athens, Athens
  - Athens Medical Center S.A - Iatriko Amarousiou, Marousi
  - Athens Medical Center- Iatriko Paleou Falirou, Palaió Fáliro
  - Geniko Nosokomeio Peiraia Tzaneio, Piraeus
  - General Hospital of Thessaloniki Ahepa, Thessaloniki
  - Thermi Clinic S.A., Thessaloniki
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Hungary (10):
  - Lausmed Kft, Baja
  - Drug Research Center Kft, Balatonfüred
  - Szent Margit Rendelointezet Diabetologiai Ambulancia, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Kft, Encs
  - Borbanya Praxis Egeszsegugyi Kft, Nyíregyháza
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft, Zalaegerszeg
- Italy (6):
  - Azienda Universitaria Ospedaliera Consorziale Policlinico Bari, Bari
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Sacco, Milan
- Japan (8):
  - Kunisaki Makoto Clinic, Fukuoka, Fukuoka
  - Nakamoto Medical Clinic, Mito, Ibaraki
  - Ohishi Naika Clinic, Tsuchiura-shi, Ibaraki
  - Morinaga Ueno Clinic, Kumamoto, Kumamoto
  - Midori Clinic, Nagasaki, Nagasaki
  - Shiraiwa Medical Clinic, Kashiwara-shi, Osaka
  - Plumeria DM Clinic, Shizuoka, Shizuoka
  - Yutenji Medical Clinic, Meguro-ku, Tokyo
- Poland (7):
  - Nzoz Specjalistyczny Osrodek Internistyczno-Diabetologiczny Malgorzata Arciszewska, Bialystok
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny numer 4 Centrum Innowacyjnych Terapii, Lublin
  - Nowe Zdrowie-Ck Kieltucki i Wspolnicy Spolka Jawna, Staszów
  - Nbr Polska Tomasz Klodawski, Warsaw
  - Centrum Badan Klinicznych Piotr Napora lekarze spolka partnerska, Wroclaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
- Latin Clinical Trial Center, San Juan, Puerto Rico
- Romania (5):
  - Mariodiab Clinic SRL, Brasov
  - Centrul pentru Studiul Metabolismului - Hightech Medical Services SRL, Bucharest
  - Institutul National de Diabet si Nutritie si Boli Metabolice N C Paulescu, Bucharest
  - Consultmed SRL, Iași
  - Clinica Korall, Satu Mare
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (5):
  - Hospital Vithas Sevilla, Castilleja de la Cuesta, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Arnau de Vilanova Lleida, Lleida, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario de La Ribera, Alzira, Valencia
- Sweden (5):
  - Ostra Sjukhuset, Gothenburg
  - Skanes universitetssjukhus, Lund
  - Universitetssjukhuset Orebro, Örebro
  - Sabbatsbergs Sjukhus, Stockholm
  - Sodersjukhuset, Stockholm
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com